CLINICAL TRIAL: NCT01847742
Title: EMDR Treatment for Psychological Trauma Among Syrian Refugees in Kilis, Randomized Controlled Trial.
Brief Title: EMDR Intervention for Psychological Trauma Among Syrian Refugees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Sehir University (Other)
Responsible Party: Principal Investigator, Ceren Acarturk, Assistant Professor, Istanbul Sehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/1No:4
Record Dates: First submitted 2013-04-21; First posted 2013-05-07 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Psychological Trauma
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMDR intervention (Experimental): 40 participants with trauma symptoms will be randomly assigned to treatment group and receive EMDR intervention for trauma symptoms.EMDR is a trauma focused therapy starts with resource development and continue with bilateral stimulation while working on the most troubling traumatic memory.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing Therapy
- Waiting List (No Intervention): 40 participants with trauma symptoms will be randomly assigned to waiting list as the control group.

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing Therapy
  Arms: EMDR intervention

SUMMARY:
To implement an EMDR (Eye Movement Desensitization and Reprocessing)intervention to treat the trauma symptoms among Syrian Refugees.

DETAILED DESCRIPTION:
In this project we aim to treat the posttraumatic stress disorder (PTSD) symptoms among Syrian refugees through an effective psycho-therapy technique called Eye Movement Desensitization and Reprocessing (EMDR). Randomly selected refugees will be assessed through MINI PLUS for the diagnose of PTSD. Eighty refugees with PTSD will be randomly allocated to either 7 sessions EMDR or wait-list control group.Symptoms of PTSD (MINI PLUS, HTQ, IES-R) and depression and anxiety (BDI, HSCL)will be assessed at pre- and post-treatment and 4 weeks follow-up.

However, to our knowledge this is one of the first intervention studies which will be conducted in a refugee camp. Therefore we expect to have some practical and logical problems. In order to see the feasibility and efficacy of EMDR among Syrian refugees, before the main study we aim to run a pilot study with less participants. In the pilot we will assess the posttraumatic stress symptoms with Impact of Event Scale-Revised (IES-R) and the depressive symptoms through Beck Depression Inventory (BDI-II).

ELIGIBILITY:
Inclusion Criteria:

* trauma symptoms

Exclusion Criteria:

* pregnancy
* current or past psychotic disorder
* current or past substance abuse or dependence
* serious physical illness
* active suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
score on Harvard Trauma Questionnaire (at the main study) | before and after the treatment,an expected average of 7 weeks of EMDR treatment
  The change in HTQ score will be assessed after the EMDR treatment has finished after 7 weeks(estimated).
Impact of Event Scale Revised (at the pilot study and the main study) | pre- and post treatment
  The change in IES-R score will be assessed after the EMDR treatment has finished after 7 weeks(estimated).

SECONDARY OUTCOMES:
score on HSCL for depressive and anxiety symptoms (at the main study) | before and after the treatment, an expected average of 7 weeks of EMDR treatment
  The change in HSCL score will be assessed after the EMDR treatment has finished in 7 weeks in average.
Score on BDI-II (pilot study and the main study) | before and after EMDR treatment, an expected average of 7 weeks of EMDR treatment
  A change in BDI-II will be assessed after the EMDR treatment has completed in 7 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Kilis Camp for Refugees, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Derived] Acarturk C, Konuk E, Cetinkaya M, Senay I, Sijbrandij M, Gulen B, Cuijpers P. The efficacy of eye movement desensitization and reprocessing for post-traumatic stress disorder and depression among Syrian refugees: results of a randomized controlled trial. Psychol Med. 2016 Sep;46(12):2583-93. doi: 10.1017/S0033291716001070. Epub 2016 Jun 29. PMID 27353367